CLINICAL TRIAL: NCT00166036
Title: Effect of Statins on Oxidative Stress and Endothelial Progenitor Cells: Comparison of Atorvastatin With Pravastatin
Brief Title: Effect of Statins on Oxidative Stress and Endothelial Progenitor Cells
Acronym: STOPCAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1038-2004
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus; Metabolic Syndrome X; Hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome; Hypercholesterolemia | interventions — Atorvastatin; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin 10MG (Experimental)
  Interventions: Drug: Atorvastatin
- Pravastatin 80mg (Experimental)
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Atorvastatin — 12 Weeks of Oral Atorvastatin 10 mg therapy.
  Arms: Atorvastatin 10MG
Drug: Pravastatin — 12 Weeks of Oral Pravastatin 80 mg therapy.
  Arms: Pravastatin 80mg

SUMMARY:
Thirty-six subjects with hyperlipidemia and metabolic syndrome and/or diabetes were randomized in a double-blind manner to either pravastatin 80 mg or atorvastatin 10 mg daily. Oxidative stress (dROMs assay that measures lipid hydroperoxides, plasma thiobarbituric acid reactive substances [TBARS], and aminothiol levels) and brachial artery flow-mediated dilation (FMD) were measured at baseline and after 12 weeks of statin therapy.

DETAILED DESCRIPTION:
Individuals with a high cholesterol level, diabetes or metabolic syndrome (collection of abnormalities such as high blood pressure, high triglyceride levels [fat], obesity, high blood glucose level) have an increased risk of developing a hardening of the arteries and heart disease.

A group of medications called statins, commonly used worldwide to lower cholesterol levels, are known to reduce the risk of heart disease through their effects on reducing cholesterol levels. These medications also have effects beyond the lowering of cholesterol that may help mediate their beneficial effects on the heart and blood vessels.

These include a reduced production of molecules that harm the arteries such as reactive oxygen species (ROS) and increasing the number of stem cells that help repair vessels, called endothelial progenitor cells (EPCs).

Recent studies have shown that different statins might have different effects on protecting people from developing heart disease. These differences may be due to differences in these non-cholesterol lowering processes, and are the subject of this study.

Standard of Care:

The two statins that will be used in this study, pravastatin (Pravachol ®) and atorvastatin (Lipitor®), are approved for use in people with a high cholesterol level or heart disease. These medications are generally very well tolerated with minimal side effects. They are not approved for use in patients to increase the level of EPCs or to reduce the production of ROS, and therefore are considered experimental for this indication. Currently there are no drugs that are specifically approved for these indications.

How the Problem Will be Studied:

These statins will be given to patients who have high cholesterol and either diabetes or the metabolic syndrome once a day for 12 weeks. We, the investigators at Emory, will measure the level of EPCs and ROS before and during the administration of the statin. We will also investigate how well the blood vessels dilate in response to these medications by performing an imaging study of the forearm artery using ultrasound.

The study is blinded and there is an equal chance of receiving either atorvastatin 10mg or pravastatin 80mg which are likely to lower cholesterol level by a similar amount.

How Research Will Advance Scientific Knowledge:

The goal of this study is to determine if atorvastatin will increase the number of circulating EPCs and reduce the production of ROS more than pravastatin. This may help explain the differences between these drugs that have been observed in some recently published trials.

ELIGIBILITY:
Inclusion Criteria:

* Males or females without child bearing potential aged 21-80 years
* Fasting low-density lipoprotein (LDL) level > 120mg/dL.
* Either known to be diabetic or have at least 3 components of metabolic syndrome that are defined below:

  * Hypertension defined as blood pressure (BP) > 140 systolic or > 90 mmHg diastolic, or stable medical therapy for documented hypertension;
  * Fasting glucose > 110 mg/dL;
  * Waist > 40 inches in males, and > 35 inches in females;
  * Triglycerides > 150mg/dL; or
  * High-density lipoprotein (HDL) cholesterol < 40 mg/dL in males and < 50 mg/dL in females.
* Able to provide written informed consent
* Non-smoker

Exclusion Criteria:

* On any oral antioxidants or lipid lowering medications in the previous 8 weeks
* Age < 21 or > 80 years
* Premenopausal females with potential for pregnancy
* LDL cholesterol level < 120 mg/dl
* Initiation or change in dose of any concomitant medical therapy within 2 months before the study
* Uncontrolled hypertension with BP > 180 mmHg systolic and > 120 mmHg diastolic
* Current smoker
* Previous intolerance or allergy to statins
* Acute infection in previous 4 weeks
* History of substance abuse
* Uninterpretable Brachial Artery Reactivity Study
* Current neoplasm
* Chronic renal failure (creatinine > 2.5 mg/dL) or liver failure (liver enzymes > 2X normal)
* Acute coronary syndrome, heart failure, cerebrovascular accident (CVA), or coronary intervention within 3 months
* Known aortic stenosis, hypertrophic cardiomyopathy, or symptomatic heart failure.
* Inability to give informed consent
* Inability to return to Emory for follow-up

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-09; Primary Completion 2008-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Murrow JR, Sher S, Ali S, Uphoff I, Patel R, Porkert M, Le NA, Jones D, Quyyumi AA. The differential effect of statins on oxidative stress and endothelial function: atorvastatin versus pravastatin. J Clin Lipidol. 2012 Jan-Feb;6(1):42-9. doi: 10.1016/j.jacl.2011.08.006. Epub 2011 Sep 13. PMID 22264573

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Previous statin or other lipid lowering medications will be discontinued for 2 months. Subjects will be on stable medical therapy for at least 2 months before recruitment.
Groups:
- Atorvastatin 10 mg; Pravastatin 80 mg: Once Daily for 12 Weeks
Period: Overall Study
Arm/Group | Atorvastatin 10 mg | Pravastatin 80 mg
Started | 17 | 19
Completed | 17 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin 10 mg: Subject treated with oral Atorvastatin 10 mg for 12 Weeks.
- Pravastatin 80 mg: Subject treated with oral Pravastatin 80 mg for 12 Weeks.
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 10 mg | Pravastatin 80 mg | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (6.6) | 51.7 (10.8) | 52.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 09 | 14 | 23
  Male | 08 | 05 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Thiobarbituric Acid Reactive Substance (TBARS) Levels
Description: Oxidative stress was assessed with plasma thiobarbituric acid reactive substance (TBARS) levels (an index of lipid peroxidation).Oxidative stress reflects an imbalance between the systemic manifestation of reactive oxygen species and a biological system's ability to readily detoxify the reactive intermediates or to repair the resulting damage.We hypothesized that equipotent doses of these two statins will have divergent effects on markers of oxidative stress and endothelial function.
Time Frame: Baseline &12 Weeks
Measure: Mean (Standard Error); unit: nmol/mL
Groups:
- Atorvastatin 10 mg: Atorvastatin 10 mg taken daily
- Pravastatin 80 mg: Pravastatin 80 mg daily
Arm/Group | Atorvastatin 10 mg | Pravastatin 80 mg
Number analyzed (Participants) | 17 | 19
nmol/mL | 2.1 (0.8) | 2.5 (1.0)

2. Secondary Outcome: Change in Flow-mediated Dilatation (FMD)
Description: Flow-mediated dilatation (FMD) of the brachial artery was used to asses Endothelial Function. The endothelium, by releasing nitric oxide (NO), promotes vasodilation and inhibits inflammation, thrombosis, and vascular smooth muscle cell proliferation.We hypothesized that equipotent doses of these two statins will have divergent effects on markers of oxidative stress and endothelial function.
Time Frame: Baseline & 12 Weeks
Measure: Mean (Standard Error); unit: Percentage of brachial artery diameter
Groups:
- Atorvastatin 10 mg: Atorvastatin 10 mg daily
Arm/Group | Atorvastatin 10 mg | Pravastatin 80 mg
Number analyzed (Participants) | 17 | 19
Percentage of brachial artery diameter | 5.9 (2.9) | 6.0 (2.3)

ADVERSE EVENTS:
Arm/Group | Atorvastatin 10 mg | Pravastatin 80 mg
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

LIMITATIONS AND CAVEATS:
Detection of changes in Oxidative stress with significance requires a much larger cohort study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No